CLINICAL TRIAL: NCT00481936
Title: A Phase I, Escalating Dose Study of VB6-845, a Recombinant Fusion Protein Targeting EpCAM, in Patients With Advanced Solid Tumours of Epithelial Origin
Brief Title: Study of the Safety of VB6-845 in Patients With Advanced Solid Tumours of Epithelial Origin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Corporate reasons unrelated to safety and efficacy
Sponsor: Sesen Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VB6-845-01-I
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Neoplasms, Glandular and Epithelial
Keywords: Neoplasms; Neoplasm, Epithelial; Neoplasm, Glandular
MeSH Terms: conditions — Neoplasms, Glandular and Epithelial; Neoplasms | interventions — VB6-845 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalating (Experimental): Patients will be treated with VB6-845 as a monotherapy IV infusion, once weekly in 4-week cycles. Patients will continue to receive treatment up until the treatment stopping criteria or patient withdrawal criteria are met.
  Dose escalation will begin at a dose level of 1.00 mg/kg. Doses will be escalated according to the modified Fibonacci design with dose multipliers of 2.00, 1.67, 1.50, 1.40, and 1.33.
  Interventions: Drug: VB6-845

INTERVENTIONS:
Drug: VB6-845 — Intravenous infusion once weekly for 4 weeks

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of VB6-845 and to evaluate the safety and tolerability of VB6-845 when administered as a monotherapy IV infusion to patients with advanced solid tumour of epithelial origin.

DETAILED DESCRIPTION:
The primary study objective of this Phase 1 trial was to determine the maximum tolerated dose (MTD) of VB6-845 and evaluate the safety and tolerability of VB6-845 when administered as a monotherapy intravenous (IV) infusion (over 3 hours), once weekly in 4-week cycles, to subjects with EpCAM positive advanced solid tumours of epithelial origin.

Secondary objectives included evaluating the pharmacokinetic profile and immunogenicity of VB6-845 and assessing exploratory efficacy of VB6-845.

Dose cohorts of 3-6 subjects with EpCAM positive advanced solid tumours of epithelial origin are to be entered into the study. The starting dose is defined as 1.00 mg/kg, which is 1/10 of the no observed adverse effect level (NOAEL) reached in preclinical studies. Doses are to be escalated according to the modified Fibonacci design until 2 out of 3 or 2 out of 6 subjects experienced a Dose Limiting Toxicity (DLT). The MTD is to be reached when <2 out of 6 subjects experienced a DLT. An additional 12 subjects are to be enrolled at the MTD for further characterization of VB6-845 at that level.

Regardless of dose cohort, subjects are to continue to receive treatment until an unacceptable toxicity occurred, all lesions completely disappeared or disease progression is determined.

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics:

* The patient must have locally advanced and/or metastatic solid tumour of epithelial origin for which standard therapy has failed or does not exist;
* The patient must have immunohistochemically-confirmed EpCAM positive disease;

Patient Characteristics:

* The patient must be male or female 18 years of age or older;
* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 and life expectancy ≥ 12 weeks
* The patient must have adequate organ function, as defined by the protocol
* Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to the first dose of the study drug;

Other:

* The patient must be able to understand and willing to sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
* The patient must be willing and able to comply with scheduled visits, the treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* The patient has had treatment with any investigational agent within 4 weeks, or treatment with radiation therapy to a visceral organ, immunotherapy, biological therapy, or chemotherapy within 2 weeks prior to the first dose of study medication
* The patient has not adequately recovered from the toxic effects of previous therapy, except treatment-related anemia otherwise meeting the inclusion requirements stated above in inclusion number 5 or alopecia;
* The patient has known clinically significant brain metastases or leptomeningeal disease (baseline computed tomography [CT] or magnetic resonance imaging [MRI] of the brain is only required if there is clinical suspicion of central nervous system involvement);
* The patient has experienced a previous significant hypersensitivity reaction;
* The patient has known acquired immune deficiency disease or has active hepatitis virus C (HVC) or active hepatitis virus B (HVB);
* The patient is pregnant or breast feeding; female patients will be required to be surgically sterile, agree to use double barrier contraception, or commit to abstinence during the period of therapy; male patients will be required to be surgically sterile, use double barrier contraception, or commit to abstinence during the period of therapy
* The patient has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness or social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of VB6-845 and to evaluate the safety and tolerability of VB6-845 when administered as a monotherapy IV infusion | 4 weeks

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics, immunogenicity and exploratory efficacy of VB6-845 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Cuthbert, Study Director — Sesen Bio, Inc.
Locations (6):
- Chemotherapy and Immunotherapy clinic Medulla, Tbilisi, Georgia
- Russia (5):
  - Blokhin Cancer Research Centre, Department of Chemotherapy and Combined therapy, Moscow
  - Blokhin Cancer Research Centre, Department of Clinical Pharmacology and Chemotherapy, Moscow
  - Moscow City Oncology Hospital #62, Moscow
  - Non state Institution of Ministry of Health "Central Clinical Hospital #2 named after N.A. Semashko" of Open-joint stock company "Russian Railways", Moscow
  - Yaroslavl Regional Clinical Oncology Hospital, Yaroslavl